CLINICAL TRIAL: NCT07382999
Title: Effect of Adherence to a Gluten-Free Diet on Cognitive and Motor Dual-Task Performance in Adolescents Diagnosed With Celiac Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Zeynal Yasacı, Doctor Lecturer, Inonu University
Other Study IDs: 1002
Record Dates: First submitted 2025-12-17; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Celiac Disease in Children; Celiac Disease in Adolescents
Keywords: Celiac; Cognitive function; 10 MWT; TMT A-B
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Celiac patients who adhere to a gluten-free diet: Patients with celiac disease who comply with the currently recognized sole treatment option-a strict gluten-free diet-will be included.
- Celiac patients who are non-compliant with a gluten-free diet: Patients with a confirmed diagnosis of celiac disease who are non-compliant with a gluten-free diet will be included.
- Healthy children without a diagnosis of celiac disease: Healthy children who have not been diagnosed with celiac disease will be included.

SUMMARY:
The aim of this cross-sectional observational study is to comprehensively examine the effects of adherence to a gluten-free diet on cognitive, motor, and psychosocial functions in adolescents aged 8-18 years diagnosed with celiac disease. In this context, dual-task gait performance, cognitive processing speed and attention, working memory and executive functions, muscle strength, quality of life, and fatigue levels of individuals with celiac disease who are adherent or non-adherent to a gluten-free diet will be compared with those of healthy peers. In addition, sleep patterns, pubertal development, socioeconomic indicators, and serological markers will be taken into account to evaluate the unique effects of diet adherence on neurocognitive and functional outcomes. All assessments will be conducted in accordance with a predefined standardized protocol. The order of measurement instruments will be randomized to minimize potential bias. Inclusion criteria will consist of being between 8 and 18 years of age, having a celiac disease diagnosis confirmed by serology, being followed with this diagnosis for at least six months, and obtaining written informed consent from both the participant and their parent/guardian. For the healthy control group, participants must be within the same age range and have no history of chronic neurological, psychiatric, or gastroenterological conditions. Data analysis will be performed using SPSS

DETAILED DESCRIPTION:
Celiac disease (CD) is an immune-mediated enteropathy triggered by the ingestion of gluten, a protein found in wheat, rye, and barley. With a global prevalence of approximately 1%, it is among the most common autoimmune disorders worldwide. Currently, the only accepted treatment is lifelong adherence to a strict gluten-free diet (GFD). It is now well recognized that CD is associated not only with varying degrees of small intestinal inflammation but also with a wide range of gastrointestinal and extraintestinal manifestations, and it may even be present in asymptomatic individuals. Common extraintestinal manifestations include abnormal liver enzymes, arthralgia/arthritis, alopecia, fatigue, headache, anemia, oral ulcers, myalgia, skin rashes, neuropathy, short stature, delayed puberty, osteoporosis, and infertility. The clinical diagnosis of CD is based on histological evaluation of small intestinal biopsies. Serological tests such as immunoglobulin A (IgA) anti-tissue transglutaminase antibodies and endomysial antibodies (EMA; IgA) may be useful in supporting the diagnosis. Several theories suggest that the globalization and spread of "incorrect" or "excessive" versions of the Mediterranean diet, characterized by very high gluten consumption (up to 20 g/day), may have contributed to the increasing prevalence and incidence of CD. In addition, gluten quality may also play a role. The production of new cereal variants for technological purposes in recent years may have influenced the observed rise in CD diagnoses. Except in regions with low frequencies of CD-predisposing genes and low gluten consumption (such as sub-Saharan Africa and Japan), CD prevalence is higher among first-degree relatives of affected individuals (10-15%) and in other high-risk groups, particularly patients with Down syndrome, type 1 diabetes, or IgA deficiency. In addition to genetic susceptibility and gluten exposure, loss of intestinal barrier function, gluten-triggered proinflammatory innate immune responses, inappropriate adaptive immune responses, and gut microbiome imbalance appear to constitute the fundamental components of CD autoimmunity. An abnormal immune response to gluten in CD classically leads to gastrointestinal symptoms such as abdominal pain, diarrhea, constipation, bloating, and weight loss. CD is now considered a multisystem disorder that affects not only the gastrointestinal tract but also the central nervous system, and has been associated with impairments in attention, short- and long-term memory, and executive function, commonly referred to as "brain fog." Dual-task (DT) gait is thought to involve higher-order cognitive processes that control and regulate behavior, including executive function, gait control, and attentional allocation. This process requires activation of multiple cortical regions, such as the prefrontal cortex (PFC), primary motor cortex, supplementary motor cortex, and somatosensory motor cortex. In addition to cortical activation, network efficiency and functional connectivity among various cortical regions, including the PFC and sensorimotor cortices, have been identified as important contributors to the cortical processes involved in DT gait. The aim of this study is to comprehensively investigate the effects of adherence to a gluten-free diet on cognitive, motor, and psychosocial functions in adolescents aged 8-18 years diagnosed with celiac disease. Accordingly, dual-task gait performance, cognitive processing speed and attentional functions, working memory and executive functions, muscle strength, quality of life, and fatigue levels of GFD-adherent and non-adherent individuals with CD will be compared with those of healthy peers. Furthermore, sleep patterns, pubertal development, socioeconomic indicators, and serological markers will be considered to evaluate the specific effects of dietary adherence on neurocognitive and functional outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged between 8 and 18 years with a serologically confirmed diagnosis of celiac disease
* Who have been followed for at least six months after diagnosisn
* For whom written informed consent has been obtained from both the participant and their parent/legal guardian, will be included in the study.
* The healthy control group will consist of individuals in the same age range with no history of chronic neurological, psychiatric, or gastroenterological diseases.

Exclusion Criteria:

* Will include the presence of an acute infection or systemic disease
* Diagnosed neurological disorders (such as epilepsy or cerebral palsy);
* A history of severe psychiatric disorders; conditions that may interfere with test administration, including visual, hearing, or ambulatory impairments
* Initiation of psychotropic medication or changes in the current dosage within the past four weeks; the presence of unstable metabolic or endocrine disorders
* Failure to obtain the required informed consent for participation.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study will include adolescents aged 8-18 years with a diagnosis of celiac disease, as well as healthy control participants from the same age group. The celiac disease group will comprise individuals who are both adherent and non-adherent to a gluten-free diet. Healthy controls will be selected from volunteers with no history of chronic neurological, psychiatric, or gastroenterological diseases.
Sampling Method: Probability Sample
Enrollment: 82 (Estimated)
Dates: Start 2026-02-12 (Estimated); Primary Completion 2026-08-15 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Dual-task 10-Meter Walk Test | baseline one assestmeant
  Following the administration of the 10-Meter Walk Test (10MWT), participants aged 6-11 years will be instructed to verbally name as many animals as they know until they are asked to stop during the test. For participants aged 12-18 years, the serial sevens task (counting backward by sevens starting from 100) will be administered concurrently with the 10MWT.

SECONDARY OUTCOMES:
10-meter walk test | Baseline one assestmeant
  A straight 10-meter walkway is used in the study; however, a 2-meter acceleration zone at the beginning and a 2-meter deceleration zone at the end of the walkway are provided. The stopwatch is started after the participant has walked the initial 2 meters and stopped before the final 2 meters. Participants are instructed to walk at their self-selected, natural, and comfortable walking speed. Walking time is recorded in seconds.
Timed Up And Go | Baseline one assestmeant
  Participants are instructed to stand up from a seated position, walk a distance of 3 meters, turn around a cone, return to the chair, and sit down again. The test performance is timed using a stopwatch and recorded in seconds.
Digit Span Test | Baseline one assestmeant
  The Digit Span Test (DST) will be administered via a mobile application, with the forward test performed by progressively increasing the sequence length. The score generated by the application will be recorded.
Trail Making Test | Baseline one assestmeant
  The mobile application version of the Trail Making Test (TMT) will be used. In Part A, numbers displayed within circles are arranged in ascending order. In Part B, both numbers and letters are presented, and participants are required to connect them in an alternating ascending sequence. Task completion time will be recorded as the outcome measure.
Tap Fast | Baseline one assestmeant
  To assess participants' reaction times, the Tap Fast mobile application will be utilized. Participants will be instructed to tap the screen as quickly as possible, touching as many targets as they can within 15 seconds. The score obtained by the participant will be recorded.
The Pediatric Quality of Life Inventory (PedsQL) | Baseline one assestmeant
  The Pediatric Quality of Life Inventory (PedsQL) will be used to assess participants' health-related quality of life. It is a brief instrument evaluating five domains: physical functioning, emotional functioning, psychosocial functioning, social functioning, and school functioning. The PedsQL is applicable to children and adolescents aged 2-18 years and includes both child self-report and parent proxy-report forms. Items are rated on a 5-point Likert scale (0-4), with higher scores indicating better quality of life.
The Pediatric Fatigue Scale | Baseline one assestmeant
  The Pediatric Fatigue Scale will be used to assess fatigue. The scale can be administered in both child self-report and parent proxy-report forms and is applicable to children and adolescents aged 2-18 years. It comprises three subscales-general fatigue, cognitive fatigue, and sleep/rest fatigue-consisting of a total of 18 items. The scale is particularly valuable for understanding the impact of chronic diseases on daily functioning and psychosocial domains. The Pediatric Fatigue Scale provides a reliable assessment of both the physical and cognitive dimensions of fatigue. Items are rated on a 5-point Likert scale (0-4), with higher scores indicating better functional capacity.
The Physical Activity Questionnaire for Children (PAQ-C) The Physical Activity Questionnaire for Adolescents (PAQ-A) | Baseline one assestmeant
  The Physical Activity Questionnaire for Children (PAQ-C) is a 9-item, 5-point Likert-type self-report measure used to assess moderate-to-vigorous physical activity levels over the previous seven days in children aged 8-14 years. The questionnaire includes items related to sports participation, school-time and out-of-school activities, physical activity during lunch breaks, and evening physical activities. Higher scores indicate better levels of physical activity.
  The Physical Activity Questionnaire for Adolescents (PAQ-A) is a 9-item, 5-point Likert-type measure designed to assess moderate-to-vigorous physical activity performed during a typical week by adolescents aged 14-18 years. While similar in structure to the PAQ-C, the PAQ-A is adapted to better reflect adolescents' daily routines, including active transportation to school, after-school activities, and weekend physical activities. Higher scores indicate better levels of physical activity.
The Pediatric Sleep Questionnaire (PSQ) | Baseline one assestmeant
  The Pediatric Sleep Questionnaire (PSQ) is used to evaluate sleep-related problems and to assess reductions in daytime functioning associated with sleep disorders. It is a parent-reported questionnaire administered to children aged 2-18 years. Section A assesses nighttime and sleep-related behaviors, Section B evaluates daytime behaviors and potential problems, and Section C consists of six items assessing attention deficit and hyperactivity symptoms. Responses to Sections A and B are recorded as "Yes," "No," or "Don't know." Items in Section C are rated on a 4-point Likert scale. For scoring purposes, responses marked as 0 or 1 are recoded as 0, whereas responses marked as 2 or 3 are recoded as 1.
  In addition, open-ended questions are included to explore the qualitative aspects of sleep problems. A total of 22 items are used in the scoring of the questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynal YASACI, Principal Investigator — İnönü Üniversitesi
Locations (1):
- İnönü Üniversitesi Turgut Özal Tıp Merkezi, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Participant data will be securely stored by the investigators and may be shared with authorized personnel if deemed necessary, in accordance with applicable privacy regulations.

REFERENCES:
- [Background] Öner P, Barut Y, Öner Ö, Üneri Ö, Bodur Ş, Turgut S, et al. [Reliability and validity of Turkish translation of the pediatric sleep questionnaire]. Klinik Psikofarmakol Bulteni. 2009;19(4):382-95.
- [Background] JANZ KF, LUTUCHY EM, WENTHE P, LEVY SM. Measuring Activity in Children and Adolescents Using Self-Report: PAQ-C and PAQ-A. Medicine & Science in Sports & Exercise. 2008;40(4):767-72.
- [Background] Varni JW, Burwinkle TM, Szer IS. The PedsQL Multidimensional Fatigue Scale in pediatric rheumatology: reliability and validity. The Journal of rheumatology. 2004;31(12):2494-500.
- [Background] Varni JW, Seid M, Kurtin PS. PedsQL™ 4.0: Reliability and Validity of the Pediatric Quality of Life Inventory™ Version 4.0 Generic Core Scales in Healthy and Patient Populations. Medical Care. 2001;39(8):800-12.
- [Background] Benton MJ, Spicher JM, Silva-Smith AL. Validity and reliability of handgrip dynamometry in older adults: A comparison of two widely used dynamometers. PLoS One. 2022;17(6):e0270132.
- [Background] Candiri B, Ramazanoglu E, Talu B, Tecellioglu M. The relationship between cognitive function and functional capacity, and cognitive reserve and reaction time in patients with multiple sclerosis. Arq Neuropsiquiatr. 2024;82(9):1-9.
- [Background] Şanlı AF, Ersöz Hüseyinsinoğlu B, Bilgiç B, Hanağası HA. Parkinson Hastalarında Algılanan ve Gerçek-Zamanlı Çift-Görev Performansının Farklı Motor-Kognitif Çift-Görev Eşleşmeleri Altında İncelenmesi. Hacettepe University Faculty of Health Sciences Journal. 2025;12(2):516-28.
- [Background] Hosoi Y, Kamimoto T, Sakai K, Yamada M, Kawakami M. Estimation of minimal detectable change in the 10-meter walking test for patients with stroke: a study stratified by gait speed. Front Neurol. 2023;14:1219505.
- [Background] Tendolkar P, Ibironke O, Marchesi G, De Luca A, Squeri V, Nolan KJ, et al. Relationship between Timed Up and Go performance and quantitative biomechanical measures of balance. Frontiers in Rehabilitation Sciences. 2024;Volume 5 - 2024.
- [Background] Ding Q, Ou Z, Yao S, Wu C, Chen J, Shen J, et al. Cortical activation and brain network efficiency during dual tasks: An fNIRS study. Neuroimage. 2024;289:120545.
- [Background] Croall ID, Tooth C, Venneri A, Poyser C, Sanders DS, Hoggard N, et al. Cognitive Impairment in Coeliac Disease with Respect to Disease Duration and Gluten-Free Diet Adherence: A Pilot Study. Nutrients. 2020;12(7).
- [Background] Caio G, Volta U, Sapone A, Leffler DA, De Giorgio R, Catassi C, et al. Celiac disease: a comprehensive current review. BMC Med. 2019;17(1):142.
- [Background] De Re V, Magris R, Cannizzaro R. New Insights into the Pathogenesis of Celiac Disease. Frontiers in Medicine. 2017;Volume 4 - 2017.
- [Background] Meyer S, Rosenblum S. Examining core self-management skills among adolescents with celiac disease. J Health Psychol. 2021;26(13):2592-602